CLINICAL TRIAL: NCT04178577
Title: A Phase 1, Open-Label Study to Assess the Pharmacokinetics and Safety of Orally Administered Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr) in Subjects With Various Degrees of Renal Function
Brief Title: Phase 1 Study of PK and Safety of Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr) in Subjects With Various Degrees Of Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPR994-102
Record Dates: First submitted 2019-11-14; First posted 2019-11-26 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2019-12

CONDITIONS: Renal Impairment
Keywords: End State Renal Disease (ESRD); Renal Insufficiency; Renal Impairment; Renal Disease; Hemodialysis
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases | interventions — tebipenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tebipenem pivoxil hydrobromide (TBPM-PI-HBr) (Experimental): Tebipenem pivoxil hydrobromide (TBPM-PI-HBr) 600 mg single-dose given orally.
  Interventions: Drug: Tebipenem pivoxil hydrobromide (TBPM-PI-HBr)

INTERVENTIONS:
Drug: Tebipenem pivoxil hydrobromide (TBPM-PI-HBr) — Tebipenem pivoxil hydrobromide (TBPM-PI-HBr) 600 mg single-dose given orally.
  Other Names: TBPM-PI-HBr; SPR994

SUMMARY:
Evaluation of the pharmacokinetics (PK) of TBPM-PI-HBr in subjects with normal renal function, subjects with various degrees of renal insufficiency, and subjects with end-stage renal disease (ESRD) receiving hemodialysis (HD) therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult males or females, 18 years of age or older.
* BMI ≥ 18.5 and ≤ 39.9 (kg/m2) and weight between 50.0 and 130.0 kg
* Medically healthy without clinically significant abnormalities (Healthy Volunteers) or medically stable without clinically significant acute or chronic illness (Subjects with Renal Disease).
* Non-smoker for at least 1 month prior to screening for the study.
* Ability and willingness to abstain from alcohol, caffeine, xanthinecontaining beverages or food.

Key Exclusion Criteria:

* Any clinically significant medical history or abnormal findings upon physical examination, or clinical laboratory tests, not specifically excluded in other criteria below that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
* Electrocardiogram (ECG) with QTcF interval duration equal or greater than 500 msec
* Hemoglobin (HB), hematocrit (HCT), white blood cell count (WBC), or platelet count less than the lower limit of normal range of the reference laboratory (Cohort 1). HB < 8.5 gm/dL, WBC ≤ 3,000 cells/μL or platelet count ≤ 100,000 cells/μL (Cohorts 2-5).
* Results of biochemistry tests for alanine aminotransferase (ALT), aspartate aminotransferase (AST) and bilirubin greater than 1.5 X the upper limit of normal (ULN) for the reference laboratory.
* Recent history of known or suspected Clostridium difficile infection.
* History of known genetic metabolism anomaly associated with carnitine deficiency (e.g., carnitine transporter defect, methylmalonic aciduria, propionic academia).
* History of chronic liver disease, cirrhosis, or biliary disease.
* History of seizure disorder except childhood history of febrile seizures.
* Positive urine drug/alcohol testing.
* Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C (HCV) antibodies.
* History of substance abuse or alcohol abuse.
* Use of antacids within 24 hours prior to study drug administration.
* Known history of clinically significant hypersensitivity reaction or anaphylaxis to any medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-09-06 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
Apparent total body clearance (CL/F). | 72 hours post dose
Area under the curve from time zero to the last quantifiable sample (AUC0-last). | 72 hours post dose
Area under the curve extrapolated to infinity (AUC0-∞). | 72 hours post dose
Apparent steadystate volume of distribution (Vss/F). | 72 hours post dose
Maximum plasma concentration (Cmax). | 72 hours post dose
Time to the maximum plasma concentration (Tmax). | 72 hours post dose
Terminal elimination half-life (t1/2). | 72 hours post dose

SECONDARY OUTCOMES:
Incidence of treatment-emergent AEs (including SAEs) categorized by severity and relationship to study drug. | 14 days post last dose
  AEs will be categorized by system organ class (SOC) and AE preferred term (PT).
Significant changes from baseline in clinical laboratory values. | 14 days post last dose
  All laboratory data will be summarized by cohort, and at each scheduled time-point using descriptive statistics (n, mean, SD, median, minimum, and maximum).
  E.g. of laboratory values: hematology, biochemistry, coagulation and urinalysis
Significant changes from baseline in physical examination. | 14 days post last dose
  Changes in baseline in physical examination findings (Normal, Abnormal NCS, Abnormal CS) will be summarized using counts and percentages by cohort, and will also be listed individually for each scheduled time-point.
  Physical examination will include: HEENT; cardiovascular, respiratory, gastrointestinal, dermatological, musculoskeletal, nervous systems, lymph nodes and general appearance. Additional body systems may be evaluated at the Investigator's discretion.
Significant changes from baseline in vitals signs. | 14 days post last dose
  Vital sign values and changes from baseline at each scheduled time-point will be summarized by cohort for the Safety Analysis Population using descriptive statistics (n, mean, SD, median, minimum, and maximum).
  Vitals signs will include: systolic and diastolic blood pressure, heart rate, respiratory rate, and temperature.
Significant changes from baseline in ECG | 14 days post last dose
  Overall evaluation of safety ECGs will be summarized by cohort, using frequency counts and percentage of subjects as normal or abnormal, and the relevance of the abnormality will be summarized by CS or NCS.
  ECG parameters will include: heart rate, RR interval, PR interval, QRS, QT and QTcF
Renal clearance (CLR) | 72 hours post dose
Fraction of drug excreted in the urine expressed as a percentage of the TBPM-PI-HBr dose administered (Ae%). | 72 hours post dose
Amount of drug excreted in the urine through 24 hours (Ae0-24), through 48 hours (Ae0-48) and through 72 hours (Ae0-72) for Cohorts 1-4. | 72 hours post dose
For subjects on dialysis, estimated hemodialysis clearance (CLHD) will be assessed. | Up to 1 day post dose - between start and end of hemodialysis.
For subjects on dialysis, the extraction ratio (ER) will be assessed. | Up to 1 day post dose - between start and end of hemodialysis.
For subjects on dialysis, the amount of the dose removed by hemodialysis (XHD) will be assessed. | Up to 1 day post dose - between start and end of hemodialysis.

OTHER OUTCOMES:
For subject in Cohort 1, cumulative amount of TBPM metabolite excreted in urine. | 72 hours post dose
For subjects in Cohort 1, cumulative urinary excretion of TBPM and TBPM metabolite as a % of dose administered. | 72 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, M.D., Study Director — Spero Therapeutics Inc
Locations (2):
- United States (2):
  - Medical Facility, Miami, Florida
  - Medical Facility, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel G, Rodvold KA, Gupta VK, Bruss J, Gasink L, Bajraktari F, Lei Y, Jain A, Srivastava P, Talley AK. Pharmacokinetics of Oral Tebipenem Pivoxil Hydrobromide in Subjects with Various Degrees of Renal Impairment. Antimicrob Agents Chemother. 2022 May 17;66(5):e0240721. doi: 10.1128/aac.02407-21. Epub 2022 Apr 14. PMID 35420493